CLINICAL TRIAL: NCT00097019
Title: A Multicenter, Single-Arm, Phase II Trial of Bevacizumab in Subjects With Platinum-Resistant Epithelial Carcinoma of the Ovary or Primary Peritoneal Carcinoma for Whom Subsequent Doxil or Topotecan Therapy Has Failed
Brief Title: A Study of Bevacizumab in Ovarian Cancer or Primary Peritoneal Cancer Where Doxil or Topotecan Therapy Has Failed
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: AVF2949g
Record Dates: First submitted 2004-11-17; First posted 2004-11-18 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Ovarian Cancer
Keywords: Recurrent ovarian cancer; Refractory ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

INTERVENTIONS:
Drug: bevacizumab

SUMMARY:
This is an open-label, single-arm, two-stage, multicenter Phase II study evaluating the efficacy and safety of bevacizumab in women with platinum resistant, advanced (Stage III or IV) EOC (epithelial ovarian cancer) or PPC (primary peritoneal cancer) that subsequently progressed either during treatment with Doxil or Hycamtin therapy or within 3 months of discontinuing treatment with Doxil or Hycamtin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Female, age >=18 years
* Advanced (Stage III or IV), histologically documented epithelial ovarian cancer or primary peritoneal cancer
* Platinum-resistant disease
* Platinum-resistant disease that subsequently progressed either during treatment with Doxil(R) or Hycamtin(R) therapy or within 3 months of discontinuing treatment with Doxil(R) or Hycamtin(R) therapy
* Received no more than three treatment regimens
* Measurable disease with at least one lesion that can be accurately measured in at least one dimension (longest dimension recorded) according to RECIST (with the exception that spiral CT scans of up to 8-mm slice thickness will be accepted)
* Recovered from prior cancer therapy (XRT, surgery, chemotherapy)
* ECOG performance status 0 or 1
* Life expectancy >12 weeks
* Use of an effective means of contraception (for women of childbearing potential)

Exclusion Criteria:

* Four or more treatment regimens
* Prior therapy with bevacizumab or other VEGF pathway-targeted therapy
* Current, recent (within 4 weeks of the first infusion of bevacizumab), or planned treatment with an experimental drug other than this Genentech-sponsored bevacizumab cancer study
* Screening clinical laboratory values: Granulocyte count <1500/uL; Platelet count <75,000/uL; Hemoglobin <8.5 g/dL (hemoglobin may be supported by transfusion or erythropoietin or other approved hematopoietic growth factors; darbopoeitin [Aranesp(R)] is permitted); Serum bilirubin >2.0 x upper limits of normal (ULN); Alkaline phosphatase, AST, and ALT >2.5 x ULN (AST, ALT >5 x ULN for subjects with liver metastasis); Serum creatinine >2.0; International normalized ratio (INR) >1.5 and activated partial thromboplastin time (aPTT) >1.5 x ULN (except for subjects receiving anticoagulation therapy); Urine protein/creatinine ratio >1.0 at screening
* Blood pressure >150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix B). Women who have received prior Doxil(R) therapy and have an ejection fraction <50% will be excluded from the study.
* History of myocardial infarction within 6 months prior to Day 0 (the day of the first bevacizumab infusion)
* History of stroke or transient ischemic attack within 6 months prior to Day 0
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0; anticipation of need for major elective surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations, or core biopsies within 7 days prior to Day 0
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Presence of central nervous system or brain metastases
* History of other malignancies within 5 years of Day 0, except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of breast, or basal or squamous cell skin cancer
* Pregnant (positive pregnancy test) or lactating
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53
Dates: Start 2005-02 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hambleton, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Result] Cannistra SA, Matulonis UA, Penson RT, Hambleton J, Dupont J, Mackey H, Douglas J, Burger RA, Armstrong D, Wenham R, McGuire W. Phase II study of bevacizumab in patients with platinum-resistant ovarian cancer or peritoneal serous cancer. J Clin Oncol. 2007 Nov 20;25(33):5180-6. doi: 10.1200/JCO.2007.12.0782. PMID 18024865